CLINICAL TRIAL: NCT04517799
Title: A Double-Blind, Crossover Trial of Cannabidiol to Treat Severe Behavior Problems in Children With Autism
Brief Title: Trial of Cannabidiol to Treat Severe Behavior Problems in Children With Autism
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Wholistic Research and Education Foundation (Unknown); Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Doris Trauner, MD, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 181455
Record Dates: First submitted 2020-08-03; First posted 2020-08-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: cannabidiol; CBD; autism; autism spectrum disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- cannabidiol (Experimental): cannabidiol arm
  Interventions: Drug: Epidiolex
- placebo (Placebo Comparator): placebo arm
  Interventions: Drug: placebo oral solution

INTERVENTIONS:
Drug: Epidiolex — While in the intervention arm subjects will receive EPIDIOLEX, an oral purified CBD solution developed by GW Pharmaceuticals. The formulation is a 100 mg/mL solution, which allows for easy dose titration and administration even to young children. EPIDIOLEX is naturally-derived CBD, and has been found to have a purity of over 98%. The solution includes a sweetener to make it palatable. Dosing is dependent upon each subject's weight.
  The dosage will be titrated over time as follows:
  Week 1: 5 mg/kg/day, divided into 2 doses Week 2: 10 mg/kg/day, divided into 2 doses Weeks 3-8: 20 mg/kg/day, divided into 2 doses If a child's weight changes by greater than 2 kg during the study, the dose will be adjusted to reflect the weight change.
  Other Names: cannabidiol
  Arms: cannabidiol
Drug: placebo oral solution — GW has developed a placebo that is identical in color and taste, and will be administered in the same volume as the CBD, so that parents and investigators should not be able to detect differences between the 2 treatments. Dosing is dependent upon each subject's weight.
  The dosage will be titrated as follows:
  Week 1: 5 mg/kg/day, divided into 2 doses Week 2: 10 mg/kg/day, divided into 2 doses Weeks 3-8: 20 mg/kg/day, divided into 2 doses If a child's weight changes by greater than 2 kg during the study, the dose will be adjusted to reflect the weight change.
  Arms: placebo

SUMMARY:
There are very few treatments that are effective in reducing severe behavioral problems associated with autism. These behaviors include aggressive and self-harm behaviors, frequent repetitive behaviors and severe hyperactivity. This study is being conducted to determine whether cannabidiol can reduce any or all of these problem behaviors.

DETAILED DESCRIPTION:
Children with autism spectrum disorders (ASD) may have severe behavior problems, including aggression, self-injurious behaviors, severe and persistent stereotypic behaviors, and extreme hyperactivity, which limit their ability to function socially and academically and are often disruptive to family life as well. Cannabidiol (CBD), a compound originally derived from the cannabis plant but without the psychoactive effects found in cannabis, has been shown to be safe and effective in the treatment of children with severe epilepsy. Two non-controlled studies using CBD from local sources have demonstrated improvements in behavior in children with autism. Parents of autistic children have been using CBD products in an unregulated fashion with unknown dosing with anecdotal reports of improved behavior. This study will use EPIDIOLEX (EPX), a purified CBD oral solution that was FDA approved in June 2018 to treat severe forms of pediatric epilepsy. Study subjects will be 30 boys between 7 and 14 years of age with autism who have severe behavior problems. Every child will undergo baseline clinical evaluation, neuropsychological, behavioral, cognitive, and language testing, will have a test of brain wave activity (EEG) and a brain MRI scan. parents will complete questionnaires on various aspects of their child's behavior. Fifteen children will receive CBD for 8 weeks and 15 will receive a placebo that looks and tastes similar to the CBD (Period 1). All of the baseline tests and questionnaires will then be repeated. After a 4 week washout period, behavioral and cognitive tests and questionnaires will be repeated and then the treatments will be reversed (Period 2). At the end of 8 weeks, all of the baseline tests and questionnaires will be repeated. Study personnel and parents will be blinded to the treatment status of each child. Statistical analyses will be used to determine whether there are significant differences between baseline testing and results after placebo or CBD treatment. Types and severities of adverse events will be tracked to provide information about the safety and tolerability of CBD in this population. If CBD is found to be safe and effective in treating the behavioral problems associated with autism, this would be a major new tool in the treatment of those children that could lead to improved functioning and quality of life for the affected individuals and their families.

ELIGIBILITY:
Inclusion Criteria:

* Boys ages 7-14 years
* Confirmed diagnosis of autism based on ADOS testing
* Autism severity assessed as severe with substantial behavioral problems

Severity of symptoms will be based on a number of criteria:

1. Aggressive and/or self-injurious (SIBs) behaviors occur almost daily (more than 6 times per week) in any situation (home, school, clinic, etc.).
2. Frequent (daily), persistent (lasting at least 5-10 minutes and repeated through the day) stereotypies (repetitive behaviors such as hand flapping, running in circles, jumping repeatedly, waving fingers in front of eyes)
3. Pervasive hyperactivity (child is so physically active that he cannot sit for meals or school work, is moving all the time, jumping off furniture, climbing onto furniture, etc.)
4. One of more of the above activities is deemed to contribute significantly to child's inability to function by parental report and with clinician agreement based on history and/or direct observation

Exclusion Criteria:

* the presence of epilepsy
* a known genetic condition such as tuberous sclerosis
* other significant health issues such as cardiac disease, presence of known congenital brain malformation, or a history of central nervous system infection.
* children who are on anticonvulsant medications such as clobazam or valproic acid will also be excluded because of potential drug-drug interactions. At the time of screening, each child's medication list will be checked for drugs that are known to cause interactions with cannabidiol.
* children with an allergy to any components of the study drug
* children who are taking CBD from another source, unless parents are willing to stop the treatment for at least 4 weeks prior to entering the study. CBD and other cannabinoid blood levels will be performed at baseline and if CBD is detected in the blood, the child will be not be included in the study.
* children who might travel out of the area for a significant time during the study
* children who recently participated in another investigational drug trial may be excluded

Ages: 7 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Score on Repetitive Behavior Scale-Revised (RBS-R) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  This scale aims to capture the frequency and severity of the repetitive and restricted behaviors that are a common feature in individuals with autism spectrum disorders. The RBS-R has been validated and has been shown to have high internal consistency and inter-rater reliability when used in outpatient settings. There are 5 subscales: Stereotypic Behavior, Self-Injurious Behavior, Compulsive Behavior, Ritualistic/Sameness Behavior, and Restricted Interests. This scale will be administered to the parent or caregiver, who will report on the child's recent behaviors. Changes in score from baseline to end of treatment will be estimated - one observed during the period of treatment with the Placebo and another during the CBD treatment - with negative value representing improvement in negative behaviors and positive value representing worsening of those characteristics.
Total Score on Child Behavior Checklist (CBCL) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  The CBCL is a widely used test that assesses problem behaviors in children by posing questions to the parent or caregiver. It poses questions about a wide range of potential negative behaviors including aggression, rule-breaking, and social problems. The school-aged scale, which will be used in this study, consists of 118 questions. The CBCL has 8 syndrome scales, including Aggressive Behavior, Anxiety/Depressed, Attention Problems, Rule-breaking, Somatic Complaints, Social Problems, Thought Problems, and Withdrawn/Depressed. Changes in score from baseline to end of treatment will be estimated - one observed during the period of treatment with the Placebo and another during the CBD treatment - with negative value representing improvement in negative behaviors and positive value representing worsening of those characteristics.
Autism Diagnostic Observation Scale- 2 (ADOS-2) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  This a widely used scale that diagnoses autism spectrum disorders across individuals with a broad range of ages, developmental levels, and language abilities. It is a semi-structured assessment and consists of behavioral observation and coding of relevant behaviors. The ADOS-2 evaluates communication, social interaction, and imaginative play. The child is asked to complete various activities and then rated on their performance by the tester. Time of administration is 40-60 minutes. Range of scores is 1-10. Changes in score from baseline to end of treatment will be estimated - one observed during the period of treatment with the Placebo and another during the CBD treatment - with negative value representing improvement in negative behaviors and positive value representing worsening of those characteristics.

SECONDARY OUTCOMES:
Total Score on Aberrant Behavior Checklist (ABC) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  This checklist relies upon parent/caregiver report to assess problematic behaviors. These behaviors are divided into 5 subscales: irritability, social withdrawal, stereotypic behavior, hyperactivity/noncompliance, and inappropriate speech.
Total Score on Social Responsiveness Scale | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  Formerly known as the Social Reciprocity Scale, this 65 item questionnaire takes a quantitative approach to measuring autistic symptomatology. It obtains "first-hand" ratings from individuals (in this case, parents) who have observed the child in naturalistic social settings. The SRS poses questions about a child's ability to engage in emotionally appropriate reciprocal social interactions, It generates a singular severity score for autistic social impairment (higher score equates with greater severity), use of which has been validated by extensive factor and cluster analyses among clinical and nonclinical populations.
Total Score on Peabody Picture Vocabulary test (PPVT-4) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  The PPVT-4 is a measure of receptive vocabulary for Standard American English. For this study we will use standard scores.
Total Score on Expressive One Word Picture Vocabulary test, Fourth Edition (EOWPVT-4) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  This test assesses the individual's ability to name a variety of objects, actions, and concepts. Participants in this study are expected to have limited verbal abilities. This test will evaluate the degree of impairment at baseline and then following treatment. Administration takes less than twenty minutes.
Total Score on Children's Sleep Habits Questionnaire (CSHQ) | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  This is a retrospective, 45-item parent questionnaire that has been used in a number of studies to examine sleep behavior in young children. Thirty-two items on the CSHQ are grouped into 8 subscales relating to a number of key sleep domains: (1) bedtime resistance (6 items); (2) sleep-onset delay (1 item); (3) sleep duration (3 items); (4) sleep anxiety (4 items); (5) night wakings (3 items); (6) parasomnias (7 items); (7) sleep-disordered breathing (2 items); and (8) daytime sleepiness (8 items). Parents are asked to recall sleep behaviors occurring during a typical recent week. A higher score is indicative of more disturbed sleep.

OTHER OUTCOMES:
Magnetic Resonance Spectroscopy | Start to finish of period 1 (8 weeks) and start to finish of period 2 (8 weeks)
  Analyses will include levels of GABA and other compounds that can be identified in MR spectra; changes in those compounds with treatment; and connectivity of different brain regions before and after treatment. MRS will examine the peaks of various neurotransmitters (glutamate, glutamine, markers of neuronal integrity (NAA) and markers of metabolic function (lactate, alanine).

CONTACTS AND LOCATIONS:
Overall Officials: Doris Trauner, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Once all data analyses have been completed, individual participant data may be available to be shared with other researchers on a case by case basis. Members of the core research team will review all requests. Data will be shared on RedCap or similar platform depending on type of data requested.

REFERENCES:
- [Derived] Trauner D, Umlauf A, Grelotti DJ, Fitzgerald R, Hannawi A, Marcotte TD, Knight C, Smith L, Paez G, Crowhurst J, Brown A, Suhandynata RT, Lund K, Menlyadiev M, Grant I. Cannabidiol (CBD) Treatment for Severe Problem Behaviors in Autistic Boys: A Randomized Clinical Trial. J Autism Dev Disord. 2025 May 24. doi: 10.1007/s10803-025-06884-y. Online ahead of print. PMID 40410546